CLINICAL TRIAL: NCT07331298
Title: Apparent Diffusion Coefficient of the Intervertebral Disc in Children: Pilot Study
Acronym: CADDIE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI19_0004 (CADDIE)
Record Dates: First submitted 2025-02-25; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Scoliosis Idiopathic
Keywords: apparent diffusion coeficient; intervertebral disc; scoliosis; child
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scoliotic patients: children with spinal deformity characterized by a hump on clinical examination and a radiological deformation in the coronal plane greater than 10 ° .
  Interventions: Other: magnetic resonance imaging of the lumbar or spinal region
- Non scoliotic patients: Childrne with no hump on clinical examination, able to walk.
  Interventions: Other: magnetic resonance imaging of the lumbar or spinal region

INTERVENTIONS:
Other: magnetic resonance imaging of the lumbar or spinal region — The duration of the acquisition sequence between 2 and 10 minutes additional compared to a conventional magnetic resonance imaging examination.

SUMMARY:
The pathophysiology of adolescent idiopathic scoliosis is unknown. This pathology develops from 10-11 years of age and progresses until skeletal maturity, or even adulthood for the most severe forms.

Current knowledge is limited as to its origin on the one hand and the evolutionary nature of scoliosis on the other.

The mechanical parameters of the intervertebral disc are incompletely known from the deep location of this organ, its fragile nature in vivo and its susceptibility to desiccation during ex-vivo analysis.

To complete our knowledge of the mechanical parameters of the intervertebral disc of scoliotic and non-scoliotic children, we are proposing an in vivo, non-invasive and non-irradiating study carried out in children who are the main target of this pathology.

The objective of this work is to characterize the diffusion parameters (apparent diffusion coefficient ADC) of the intervertebral disc in vivo, in a non-invasive and non-irradiating manner by magnetic resonance imaging in children and adolescents. As this measurement has not been carried out in children and adolescents, we want to perform these MRI scans in children free from scoliosis and carriers of scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* age: patients between 8 and 16 years old
* Children undergoing magnetic resonance imaging of the lumbar or spinal region as part of their routine care
* Scoliotic: spinal deformity characterized by a hump on clinical examination and a radiological deformation in the coronal plane greater than 10 ° with no etiology found (idiopathic)
* Healthy: no hump on clinical examination, walking patients (level 1 and 2 of the global motor function classification system)

Exclusion Criteria:

* existence of medullary and vertebral pathology other than scoliosis, history of disc or vertebral infection (spondylo-discitis) on examination, neuro-ectodermal pathology
* behavioral disturbances incompatible with the performance of the magnetic resonance imaging examination.
* Refusal of participation.
* Thoracic scoliosis

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children and adolescents with and without scoliosis seen in consultation and requiring magnetic resonance imaging of the lumbar region
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
measurement of the value of Apparent Diffusion Coefficient (ADC) in magnetic resonance imaging. | between Day 15 and Day 90

SECONDARY OUTCOMES:
Apparent Diffusion Coefficient difference for scoliosis and non-scoliosis patients for one level | between Day 15 and Day 90
Correlation between right and left Apparent Diffusion Coefficient and inclination of two vertebra for scoliosis patients | between Day 15 and Day 90
gagCEST(Chemical Exchange Saturation Transfer) measurement in magnetic resonance imaging of the discs | between Day 15 and Day 90

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Limoges University Hospital, Limoges
  - Toulouse University Hospital, Toulouse